CLINICAL TRIAL: NCT02903199
Title: The Effect of Pre-meal Whey Protein on Glycaemic and Appetite Responses in Type II Diabetic Males
Brief Title: Whey Protein Effect on Glycaemic and Appetite Responses in T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NorthumbriaT2D
Record Dates: First submitted 2016-08-02; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Type II Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases
Keywords: Whey Protein; Postprandial Glycaemia; Appetite Response
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whey Protein (Experimental): Whey protein (18g) experimental supplement
  Interventions: Dietary Supplement: Whey Protein
- Hydrolysed Protein (Experimental): Hydrolysed whey protein (19.1g) experimental supplement
  Interventions: Dietary Supplement: Hydrolysed Protein
- Placebo (Placebo Comparator): Water placebo supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey Protein — Whey protein (18 g) administered immediately prior to breakfast and lunch meals.
  Arms: Whey Protein
Dietary Supplement: Hydrolysed Protein — Hydrolysed whey protein (19.1 g) administered immediately prior to breakfast and lunch meals.
  Arms: Hydrolysed Protein
Dietary Supplement: Placebo — Placebo intervention administered immediately prior to breakfast and lunch meals.
  Arms: Placebo

SUMMARY:
The current study will investigate the effect if whey protein on postprandial glycaemia and appetite in type II diabetics, assessing incretin (GLP-1, GIP), insulin, and appetite control (leptin, PYY3-36) hormone responses.

DETAILED DESCRIPTION:
Whey protein accounts of ~20% of whole milk protein. Ingestion of whey protein at meal times generates insulinotrophic/β-cell stimulation via amino acid absorption and the bioactive peptides generated during gastrointestinal digestion, resulting in attenuation of postprandial blood glucose. The bioactive peptides stimulate the release of incretin hormone, GLP-1, and inhibit DPP-IV activity potentially decreasing the rate of GLP-1 degradation.

The current study will employ a randomised, double-blind, counter-balanced, cross-over design, whereby participants will each complete three trials; a) whey protein, b) hydrolysed protein, and c) placebo intervention. Hydrolysed protein provides amino acid content, without bioactive peptides associated with incretin release, therefore, demonstrating insulinotrophic properties, only.

Many studies within the literature are limited for practical reasons, such as investigating high dosages (30-50 g) of whey protein, or high glycaemic index meal types which would be unlikely to form part of habitual dietary activity of type II diabetics. Therefore, the current study will objectively measure postprandial glycaemic and appetite responses following the ingestion of whey/hydrolysed protein, whilst ensuring ecological validity, dosages (18 g) and test meals applicable to everyday life, and true clinical utility for managing type-II diabetes by integrating interventions into the habitual lives of type-II diabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetic males aged 18-65 years old.
* Treated with metformin, or diet and lifestyle modification, only.
* BMI < 40 kg/m2.
* Stable physical activity pattern during the three months immediately preceding study.

Exclusion Criteria:

* Not treated with insulin.
* No metabolic disease other than diabetes.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Postprandial capillary glucose | 6 hours per week, for 3 weeks.
  Capillary glucose concentrations are monitored for 6 hours/wk following breakfast (09:00-12:00) and lunch (12:15-15:15).

SECONDARY OUTCOMES:
Plasma Glucagon-like Peptide-1 (GLP-1) | 3 weeks
  GLP-1 will be measured from blood collection tubes containing EDTA, aprotinin, and DPPIV inhibitor.
Plasma Gastric Inhibitory Polypeptide (GIP) | 3 weeks
  GIP will be measured from blood collection tubes containing EDTA, aprotinin, and DPPIV inhibitor.
Plasma Leptin | 3 weeks
  Leptin will be measured from blood collection tubes containing EDTA, aprotinin, and DPPIV inhibitor.
Plasma Peptide YY (PYY3-36) | 3 weeks
  PYY3-36 will be measured from blood collection tubes containing EDTA, aprotinin, and DPPIV inhibitor.
Plasma Insulin | 3 weeks
  Insulin will be measured from blood collection tubes containing EDTA, aprotinin, and DPPIV inhibitor.
Serum Triglycerides | 3 weeks
  Triglycerides will be measured from Serum Separating Tubes (SST).
Serum Glycerol | 3 weeks
  Glycerol will be measured from Serum Separating Tubes (SST).
Self-Report Questionnaire for Appetite | 3 weeks
  Visual Analogue Scales (VAS) will be used to assess self reported feelings of appetite sensations (i.e. hunger, satiety, prospective food intake).
24 h Interstitial Glucose | 3 days per week, for 3 weeks
  Interstitial glucose is measured from 36 h prior to the trial, until 24 h following the trial, each week for three weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Walker, Principal Investigator — Newcastle University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] King DG, Walker M, Campbell MD, Breen L, Stevenson EJ, West DJ. A small dose of whey protein co-ingested with mixed-macronutrient breakfast and lunch meals improves postprandial glycemia and suppresses appetite in men with type 2 diabetes: a randomized controlled trial. Am J Clin Nutr. 2018 Apr 1;107(4):550-557. doi: 10.1093/ajcn/nqy019. PMID 29635505